CLINICAL TRIAL: NCT07377565
Title: A First-in-Patient Study to Evaluate the Safety and Tolerability of HB-2121 as a Diagnostic for Celiac Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nielsen Fernandez-Becker (Other)
Collaborators: Stanford's Innovative Medicines Accelerator (Unknown)
Responsible Party: Sponsor-Investigator, Nielsen Fernandez-Becker, Clinical Professor, Medicine - Gastroenterology & Hepatology, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pending
Record Dates: First submitted 2026-01-09; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-07

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; HB-2121; Gluten Intolerance; Esophagogastroduodenoscopy
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 250 mg HB-2121 in Participants with Suspected Celiac Disease (Experimental): Participants in this arm will receive a one-time dose of 250 mg of HB-2121.
  Interventions: Drug: HB-2121

INTERVENTIONS:
Drug: HB-2121 — HB-2121 taken once orally.

SUMMARY:
The goal of this clinical trial is to learn about the safety of a single dose of HB-2121 in adults with suspected celiac disease. It will also look at how the drug affects the small intestine. The main questions it aims to answer are:

* What side effects do participants have after receiving HB-2121?
* How does the drug interact with the small intestine in people with suspected celiac disease?

Researchers will follow participants for 30 days after receiving HB-2121 to understand how the drug behaves in the body and how safe it is.

Participants will:

* Receive one oral dose of HB-2121 four hours before their standard-of-care esophagogastroduodenoscopy
* Attend 4 in-person clinic visits for checkups, lab tests, and monitoring
* Complete 2 remote visits that include safety lab assessments
* Fill out a short daily questionnaire for 7 days about symptoms and health status

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years
* Undergoing esophagogastroduodenoscopy (EGD) for suspected celiac disease
* Body Mass Index (BMI) between 18 and 45 kg/m2
* Creatinine <1.5 x Upper Limit of the Normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL x (ULN)
* Aspartate aminotransferase (AST)/Serum glutamic oxaloacetic transaminase (SGOT) & Alanine Aminotransferase (ALT)/Serum glutamic pyruvic transaminase (SGPT) ≤ 1.5 x ULN
* Overall good health, as determined by medical history and a physical exam
* No use of an investigational drug within 12 weeks
* Able and willing to follow study procedures and provide written informed consent
* If of childbearing potential, participants must agree to use highly effective birth control during the study period. The same applies to male participants with partners of childbearing potential

Exclusion Criteria:

* Pregnant, breastfeeding, planning to become pregnant, or intending to donate eggs during the study period
* History of cancer or malignancy
* History of chemotherapy and/or pelvic radiation
* History of congenital long QT syndrome or prolonged QTcF interval
* Prisoners, institutionalized individuals, or individuals who are unable to consent for themselves
* Known HIV infection, or positive test for hepatitis B or C, or other clinically significant chronic liver disease
* Current use of immunosuppressant medications
* Known allergy or sensitivity to any ingredients in the study drug
* History of eosinophilic enteritis, Crohn's disease, or ulcerative colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events during the study window | From dosing through 30 days post-dose
  Adverse events (AEs) will be recorded and assessed for severity using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Intensity of sulfo-Cy5 fluorescent marker normalized to the mean fluorescence intensity of DAPI-stained nuclei in a confocal fluorescent microscopic field of view. | 240 minutes after dosing
  Endoscopic biopsy samples will be collected after dosing, and fresh frozen tissue sections will be stained with DAPI and analyzed using a confocal microscope to determine the fluorescence intensity of sulfo-Cy5 and DAPI.
Measurement of villous height to crypt depth ratio and intraepithelial lymphocyte count. | 240 minutes after dosing
  Endoscopic biopsy samples will be collected after dosing, and the paraffin-embedded tissue sections will be stained with hematoxylin and eosin, as well as CD3, and analyzed using a microscope to determine villus height, crypt depth, and the number of CD3+ intraepithelial lymphocytes.

OTHER OUTCOMES:
Frequency and identity of HB-2121 positive cells in the blood of celiac patients | Pre-dose and at 360 minutes after dosing
  Blood samples will be collected at the end of the overall endoscopic evaluation procedure, and peripheral blood mononuclear cells (PBMCs) will be analyzed using flow cytometry to determine the percentage of HB-2121+ cells among CD14+CD11c+ populations, with and without β7-integrin expression.
Intensity of of HB-2121-labeled ECM-associated and cellular TG2 protein in duodenal biopsy samples. | 240 minutes after dosing
  Endoscopic biopsy samples will be collected after dosing, and the paraffin-embedded tissue sections will be stained with Collagen 1, PDGFRα, αSMA, CD11c, as well as DAPI, and analyzed using the confocal microscope to determine HB-2121 colocalization with ECM proteins and cell populations.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Medicine Clinical and Translational Research Unit (CTRU), Palo Alto, California, United States